CLINICAL TRIAL: NCT03918460
Title: Treatment of Type II Endoleak With ANEUFIX: Assessment of Safety, Performance and Clinical Benefit.
Brief Title: ANEUFIX for Endoleak Type II Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TripleMed B.V. (Industry)
Collaborators: Trium Clinical Consulting (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TripleMed 002
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Abdominal Aortic Aneurysm; Endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Intervention Model Description: The current study is a follow up study on the previous feasibility study where ACP-T5 was used; after increasing the % tantalum in ANEUFIX to make the product more detectable under X-ray, the current study evaluates the end-points in a total of 40 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All patients enrolled are intended to be treated
  Interventions: Device: ANEUFIX

INTERVENTIONS:
Device: ANEUFIX — ANEUFIX is administered through translumbar injection into the AAA using imaging techniques to guide the place of injection.

SUMMARY:
The study is non-randomized, multicenter international safety, performance and clinical benefit outcome assessment of ANEUFIX to treat patients with isolated type II endoleak in the presence of a growing AAA-sac following an EVAR procedure more than 6 months ago.

DETAILED DESCRIPTION:
The investigational device is called ANEUFIX, which is a product treating the endoleak by blockage of backflowing blood vessels, i.e. by filling the endoleak void and nidus of feeding artery and exit of existing draining arteries.

ANEUFIX is a polymer that cures rapidly (2-4 min at 37°C) after injection into the AAA-sac close to the nidus.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent type II endoleak (more than 6 months post-EVAR or post-embolization procedure); AND
2. An endoleak confirmed on a CT scan that should be done within 180 days prior to procedure but preferably within 90 days prior to screening demonstrating the high likelihood of the isolated nature of the endoleak; AND
3. An aneurysm sac growing after EVAR of minimal 10 mm (per European Guidelines) as documented in the preceding 90 days by means of CT-imaging (or alternative imaging techniques) and based upon sac diameter measurements; AND
4. An aneurysm sac that can be punctured via a translumbar approach; AND
5. Possibility to withhold anti-thrombogenic medication temporarily; AND
6. Ability and willingness to undergo the translumbar procedure; AND
7. Being older than 18 years.

Exclusion Criteria:

1. Patient not able or willing to give written Informed Consent; OR
2. Patient undergoing emergency procedures; OR
3. Patient with traumatic vascular injury; OR
4. Patient with haemostatic disorder (including bleeding disorders) or who is clinically unstable; OR
5. Patient with a too high risk of abdominal sac rupture to allow safe radiological and scanographic assessments; OR
6. Patient who is allergic to contrast media or anticoagulants; OR
7. Patient with renal impairment (eGFR < 30 ml/min); OR
8. Patient with a contra-indication for temporal positioning of a translumbar needle/catheter; OR
9. Patient who is participating in another trial with an investigational drug or medical device, or where a medical device/drug is used outside its labelling and its approved intended use; OR
10. Pre-menopausal women, OR
11. Patient with a life expectancy of less than 12 months, OR
12. Patient with an intra aneurysm systolic blood pressure > 125 mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | 24 hours
  Technical success of Type II endoleak repair with Aneufix as demonstrated by the absence of endoleak circulation at the intended treated endoleak at the end of the procedure; presence or absence of the endoleak treated with ANEUFIX is verified by means of a CT scan the next day.

SECONDARY OUTCOMES:
Absence of aneurysm sac growth | 6, 12 and 14 months
  Absence of aneurysm sac growth at 6, 12 and 24 months. Growth is determined based on independent core lab assessments of the abdominal aortic diameter, measured as the maximum diameter relative to the aneurysm.
Intra- and peri-operative complications | 30 days
  Documentation of intra- and peri-operative complications
serious adverse events, vascular related adverse events and adverse device effects: complications and deaths, re-interventions, aneurysm rupture | During the Aneufix procedure
  Occurrence of serious adverse events, vascular related adverse events and adverse device effects: complications and deaths, re-interventions, aneurysm rupture in the peri operative period.
Occurrence of general adverse events and adverse device effects | 1 week and 1, 6, 12 and 24 months
  Safety is assessed based on the nature and severity of observed adverse events
Rate of re-interventions | 1, 6, 12 and 24 months
  Rate of secondary endovascular or surgical re-interventions
Rate of aneurysm rupture | 6,12 and 24 months
  Rate of aneurysm rupture will be observed
Survival rate | 24 months
  Survival throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Arjan WJ Hoksbergen, Dr, Principal Investigator — VUmc Heelkunde, Amsterdam
Locations (9):
- Belgium (3):
  - Imelda, Bonheiden
  - ZOL, Genk
  - UZ Leuven, Leuven
- Netherlands (6):
  - ZGT, Almelo
  - Amsterdam UMC - VUmc, Amsterdam
  - OLVG, Amsterdam
  - Rijnstate, Arnhem
  - Spaarne Gasthuis, Haarlem
  - ETZ, Tilburg

IPD SHARING:
Plan to Share IPD: No